CLINICAL TRIAL: NCT04435470
Title: Epidemiological Study of the Microbiota in Critically Ill Children and Its Relationship With Clinical Complications and Inflammation Biomarkers
Brief Title: Epidemiological Study of the Microbiota in Critically Ill Children
Acronym: BIOUCIP
Status: Completed | Type: Observational
Sponsor: Universidad de Granada (Other)
Collaborators: Hospital Materno-Infantil Torrecárdenas de Almería (Unknown); Hospital Materno-Infantil de Málaga (Other); Complejo Hospitalario Universitario de Santiago (Other); University Hospital Virgen de las Nieves (Other)
Responsible Party: Principal Investigator, María Dolores Mesa García, Associate Professor, Universidad de Granada
Other Study IDs: BIOUCIP; PI18/01334 (Other Grant/Funding Number: Proyectos de Investigación en Salud ISCIII Spain)
Record Dates: First submitted 2020-06-11; First posted 2020-06-17 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Critical Illness; Child, Only; Intensive Care Unit
Keywords: microbiota; inflammation; metabolomic
MeSH Terms: conditions — Critical Illness; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma Feces Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Critical ill children: Critial ill children admited in pediatric intensive care units 1-16 years old
- Control: Healthy children 1-16 years old

SUMMARY:
Objectives: To study the composition of the microbiota in critically ill children, and to know the relationship of its microbiota with clinical complications and inflammation biomarkers.

Design: Multicenter observational and prospective study including 100 critically ill children admitted in three pediatric intensive care units with a prediction of more than 5 days of stay and 50 healthy children. Clinical parameters and rectal, fecal, blood and respiratory samples will be collected at admission and at pediatric intensive care units discharge. The microbiota and inflammation biomarkers and metabolomic will be analyzed.

Analysis of results: Description an evolution of the microbiota throughout the time, intestinal and respiratory, and the influence of clinical and therapeutic factors will be analyzed. The composition of microbiota will be compared with a cohort of healthy children and between the different types of pediatric intensive care units. The correlation of the microbiota with the markers of inflammation, metabolomics and the development of infectious complications and multiorgan failure will be analyzed.

DETAILED DESCRIPTION:
AIM: The present study is an observational clinical study aimed to study the intestinal microbiota composition of critically ill children in paediatric intensive care unit and its relationship with clinical complications and inflammatory biomarkers.

DESIGN: This study is a multicentre, observational and prospective study including 100 critically ill children admitted in three paediatric intensive care units (Hospital Materno-Infantil Torrecárdenas de Almería, y en el Hospital Materno-Infantil Carlos Haya de Málaga and Complejo Hospitalario Universitario de Santiago) This study is a multicentre, observational and prospective study conducted by members of the Department of Biochemistry and Molecular Biology II, Nutrition and Food Technology Institute "José Mataix" of the University of Granada research group in collaboration with the Hospital Materno-Infantil Torrecárdenas from Almería, the Hospital Materno-Infantil Carlos Haya from Málaga and Complejo Hospitalario Universitario from Santiago de Compostela pediatric intensive care units and primary care unit of the University Hospital Virgen de las Nieves from Granada as recruitment centres.

This trial will include 100 critically ill children admitted from the three different pediatric intensive care units with an expected hospitalization time of more than 5 days. In addition, 50 healthy children will be recruited from a primary care centre as controls. Faecal and respiratory system (oropharynx) samples will be collected from ill and healthy children, while blood samples will be harvested only from critically ill children at the time of admission to the pediatric intensive care units as well as at the day of discharge. Sample aliquots will be sent to the Department of Biochemistry and Molecular Biology II, University of Granada for further analysis.

Study population The study population will comprise 50 healthy children aged between 1 month and 16 years, recruited in a paediatric primary care center from Granada, and 100 critically ill children admitted to the pediatric intensive care units aged between 1 month and 16 years. 50 patients will be recruited at the pediatric intensive care units of Hospital Materno-Infantil Torrecárdenas from Almería, the Hospital Materno-Infantil Carlos Haya from Málaga and Complejo Hospitalario Universitario from Santiago de Compostela. Only those children who satisfy all inclusion and none of exclusion criteria will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* admission to pediatric intensive care unit
* hospitalization time expectancy more than 5 days
* age between 1 month and 16 years
* informed consent signed

Exclusion Criteria:

* hospitalization time expectancy less than 5 days
* no signed informed consent

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Critical ill children admited to pediatric intensive care unit, with a hospitalization time expectancy more than 5 days Control subjects will be healthy children
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
To identify intestinal and respiratory microbiota and if their changes are related with digestive and infectious complications | At admission and through study completion, at least 5 days
  To analyse the intestinal and respiratory microbiota in critically ill children admitted to the pediatric intensive care unit through massive sequencing, and evaluate if their changes are related with the appearance of digestive and infectious complications and the development of multiorgan failure.

SECONDARY OUTCOMES:
To compare intestinal and respiratory microbiota of critically ill children with a cohort of healthy children | Samples will be taken at admission to pediatric intensive care unit and a single sample witl be taken from healthy controls
  To compare intestinal and respiratory microbiota of critically ill children when admitted to the pediatric intensive care unit with a cohort of healthy children
To study the clinical factors influencing the changes in the intestinal microbiota during admission to the pediatric intensive care unit | At admission and through study completion, at least 5 days
  To study the clinical factors and influencing the changes in the intestinal microbiota during admission to the pediatric intensive care unit
To compare the changes of the microbiota according to the type of critical patients and the type of pediatric intensive care unit | At admission and through study completion, at least 5 days
  To compare the changes in the composition of intestinal and respiratory microbiota according to the type of critical patients and the type of pediatric intensive care unit
To assess the relationship between changes in the intestinal microbiota and the frequency and severity of digestive complications | At admission and through study completion, at least 5 days
  To assess the relationship between the composition of the intestinal microbiota and the frequency and severity of digestive complications (diarrhea, constipation and tolerance of enteral nutrition) in critical ill children admitted to the pediatric intensive care unit
To study the relationship between changes in the intestinal and respiratory microbiota and the frequency and severity of nosocomial infection | At admission and through study completion, at least 5 days
  To study the relationship between the composition of intestinal and respiratory microbiota and the frequency and severity of nosocomial infection in critically ill children admitted to the pediatric intensive care unit
To study the relationship between changes in the intestinal and respiratory microbiota and the development of multiorgan failure | At admission and through study completion, at least 5 days
  To study the relationship between the intestinal and respiratory microbiota and the development of multiorgan failure in critical ill children admitted to the pediatric intensive care unit
To determine changes in the serum levels of lipopolysaccharide and lipopolysaccharide binding protein and to evaluate their relationship with intestinal and respiratory microbiota | At admission and through study completion, at least 5 days
  To determine the serum levels of lipopolysaccharide (LPS) and lipopolysacchaide binding protein (LPB) in critical ill children admitted to the pediatric intensive care unit, and to evaluate their relationship with intestinal and respiratory microbiota, the evolution during admission and the relationship with clinical complications
To analyse the relationship between changes in the intestinal and respiratory microbiota plasma sort chain fatty acids and bile acids | At admission and through study completion, at least 5 days
  To analyse the relationship between the intestinal and respiratory microbiota and the metabolomic profile, especially short chain fatty acids (SCFA) and bile acids, in critical ill children admitted to the pediatric intensive care unit, the evolution during admission and the relationship with clinical complications
To analyse the relationship between changes in microbiota and inflammatory biomarkers | At admission and through study completion, at least 5 days
  To analyse the relationship between microbiota and inflammatory biomarkers in critical ill children admitted to the pediatric intensive care unit, the evolution during admission and the relationship with clinical complications
To assess the influence of the type of nutrition during admission and changes of intestinal microbiota | At admission and through study completion, at least 5 days
  To assess whether the type of nutrition, enteral or parenteral, of critical ill children during admision to pediatric intensive care unit and to evaluate their influences with the composition of the intestinal microbiota, and the relationship with clinical complications

CONTACTS AND LOCATIONS:
Overall Officials: MARÍA DOLORES MESA GARCÍA, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- María Dolores Mesa García, Armilla, Granada, Spain

IPD SHARING:
Plan to Share IPD: No
Study Protocol